CLINICAL TRIAL: NCT03944135
Title: Effectiveness of Two Predefined Groups With Cognitive Rehabilitation in Older Adults With the Program Neuron-up
Brief Title: Cognitive Rehabilitation in Older Adults With Neuron-up (CROAN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UBurgos; IR 10/2019 (Registry Identifier: UBurgos)
Record Dates: First submitted 2019-03-11; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Indication for Modification of Patient Cognitive Status
Keywords: Cognition, Cognitive Dissonance, Geriatrics, Technology

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental design with non-equivalent groups (pretest-posttest) carried out in a more realistic setting, where the dependent variables of interest were manipulated by the researcher under controlled conditions.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The sample consisted of 40 people: 20 in an experimental group. There were 5 men and 15 women.
  Interventions: Other: Web platform: Neuronup
- Control group (Active Comparator): The sample consisted of 40 people: 20 in a control group. There were 5 men and 15 women.
  Interventions: Other: Web platform: Neuronup

INTERVENTIONS:
Other: Web platform: Neuronup — Neuronup is a web platform designed for neuropsychological rehabilitation that is focused on functional cognitive impairments resulting from normal aging and other causes. Neuronup emerged as a scientific, viable and accessible technological initiative.

SUMMARY:
Introduction. The application of new technologies for cognitive rehabilitation has increased over the last years and has enabled occupational therapists to work more efficiently, minimizing costs and time for analysis, management, and design of activities.

Objective. The purpose of the present study was to assess the effect of cognitive intervention using the web platform Neuronup in a group of elderly subjects; the study is based on the dependent variables (memory, attention, and language) analyzed with the abbreviated Barcelona Test.

Subjects and Methods. Aquasi-experimental design was carried out with subjects assigned to two groups: a control group (20 subjects) and an experimental group (20 subjects). The abbreviated Barcelona Test was administered to assess patients before and after the intervention with this software to draw conclusions.

DETAILED DESCRIPTION:
Introduction. The application of new technologies for cognitive rehabilitation has increased over the last years and has enabled occupational therapists to work more efficiently, minimizing costs and time for analysis, management, and design of activities.

Objective. The purpose of the present study was to assess the effect of cognitive intervention using the web platform Neuronup in a group of elderly subjects; the study is based on the dependent variables (memory, attention, and language) analyzed with the abbreviated Barcelona Test.

Subjects and Methods. Aquasi-experimental design was carried out with subjects assigned to two groups: a control group (20 subjects) and an experimental group (20 subjects). The abbreviated Barcelona Test was administered to assess patients before and after the intervention with this software to draw conclusions.

Results. Analyses of variance (ANOVA), analyses of covariance (ANCOVA), and multivariate analyses of variance (MANOVA) were perfomed in the memory, orientation, reading, and language domains. Statistically signifcant differences were recorded in all domains except language where scores remained the same.

Conclusion. It has been demonstrated that Neuronup is an effective program for improving cognitive processes such as memory, attention, and orientation in older adults, hence it would be beneficial to implement technology-based treatments conducted by specialized professionals.

ELIGIBILITY:
Inclusion Criteria:

1. subjects between 75 and 85 years of age;
2. obtain a score greater than 20 points for the MEC (Lobo's cognitive mini-exam); and
3. attend occupational therapy sessions on a regular basis.

Exclusion Criteria:

1. presence of neurocognitive disorder (Alzheimer's-type dementia among others);
2. not be an institutionalized resident at a nursing home;
3. a family history of a psychiatric problem;
4. presence of polipathology; and
5. have lived at a nursing home for less than 2 months.

Ages: 75 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Reading is assessed in two pre defined groups of individuals | 3 months
  The abbreviated Barcelona Test is used to assess cognitive reading function in which the results highlight the existence of statistically significant differences in the difference scores reading.
  The test consists of 41 subtests that generate 55 variables which assess the following cognitive functions: language, orientation, forward/backward digit span, automatized sequences and mental control, repetition, confrontation naming, semantic fluency (animals), verbal comprehension, reading, writing, praxis (ideomotor, melokinetic, and constructional), visual perceptual functions, verbal memory (story), visual memory, arithmetic problems, similarities, digit-symbol and block design. The cognitive profile and global scale score were obtained from all scores.
Memory is assessed in two pre defined groups of individuals | 3 months
  The abbreviated Barcelona Test is used to assess cognitive memory function in which the results highlight the existence of statistically significant differences in the difference scores memory.
  The test consists of 41 subtests that generate 55 variables which assess the following cognitive functions: language, orientation, forward/backward digit span, automatized sequences and mental control, repetition, confrontation naming, semantic fluency (animals), verbal comprehension, reading, writing, praxis (ideomotor, melokinetic, and constructional), visual perceptual functions, verbal memory (story), visual memory, arithmetic problems, similarities, digit-symbol and block design. The cognitive profile and global scale score were obtained from all scores.
Orientation is assessed in two pre defined groups of individuals | 3 months
  The abbreviated Barcelona Test is used to assess cognitive orientation function in which the results highlight the existence of statistically significant differences in the difference scores orientation.
  The test consists of 41 subtests that generate 55 variables which assess the following cognitive functions: language, orientation, forward/backward digit span, automatized sequences and mental control, repetition, confrontation naming, semantic fluency (animals), verbal comprehension, reading, writing, praxis (ideomotor, melokinetic, and constructional), visual perceptual functions, verbal memory (story), visual memory, arithmetic problems, similarities, digit-symbol and block design. The cognitive profile and global scale score were obtained from all scores.

CONTACTS AND LOCATIONS:
Overall Officials: Olalla Saiz Vazquez, Principal Investigator — Universidad de Burgos
Locations (1):
- Olalla Saiz Vazquez, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohs RC, Ashman TA, Jantzen K, Albert M, Brandt J, Gordon B, Rasmusson X, Grossman M, Jacobs D, Stern Y. A study of the efficacy of a comprehensive memory enhancement program in healthy elderly persons. Psychiatry Res. 1998 Feb 27;77(3):183-95. doi: 10.1016/s0165-1781(98)00003-1. PMID 9707301
- [Background] Dellefield KS, McDougall GJ. Increasing metamemory in older adults. Nurs Res. 1996 Sep-Oct;45(5):284-90. doi: 10.1097/00006199-199609000-00006. PMID 8831655
- [Background] Wilkinson AJ, Yang L. Long-Term Maintenance of Inhibition Training Effects in Older Adults: 1- and 3-Year Follow-Up. J Gerontol B Psychol Sci Soc Sci. 2016 Jul;71(4):622-9. doi: 10.1093/geronb/gbu179. Epub 2015 Jan 7. PMID 25573153
- [Background] Neely AS, Backman L. Effects of multifactorial memory training in old age: generalizability across tasks and individuals. J Gerontol B Psychol Sci Soc Sci. 1995 May;50(3):P134-40. doi: 10.1093/geronb/50b.3.p134. PMID 7767691
- [Background] Lachman ME, Weaver SL, Bandura M, Elliott E, Lewkowicz CJ. Improving memory and control beliefs through cognitive restructuring and self-generated strategies. J Gerontol. 1992 Sep;47(5):P293-9. doi: 10.1093/geronj/47.5.p293. PMID 1512434
- [Background] Valentijn SA, van Hooren SA, Bosma H, Touw DM, Jolles J, van Boxtel MP, Ponds RW. The effect of two types of memory training on subjective and objective memory performance in healthy individuals aged 55 years and older: a randomized controlled trial. Patient Educ Couns. 2005 Apr;57(1):106-14. doi: 10.1016/j.pec.2004.05.002. PMID 15797159
- [Background] Floyd M, Scogin F. Effects of memory training on the subjective memory functioning and mental health of older adults: a meta-analysis. Psychol Aging. 1997 Mar;12(1):150-61. doi: 10.1037//0882-7974.12.1.150. PMID 9100276
- [Background] Valencia C, Lopez-Alzate E, Tirado V, Zea-Herrera MD, Lopera F, Rupprecht R, Oswald WD. [Cognitive effects of combined memory and psychomotor training in elderly adults]. Rev Neurol. 2008 Apr 16-30;46(8):465-71. Spanish. PMID 18428103
- [Background] E Mintzer J, F Mirski D, S Hoernig K. Behavioral and psychological signs and symptoms of dementia: a practicing psychiatrist's viewpoint. Dialogues Clin Neurosci. 2000 Jun;2(2):139-55. doi: 10.31887/DCNS.2000.2.2/jmintzer. PMID 22034243
- [Background] Valdizan JR. [Cognitive functions and neuronal networks in the social brain]. Rev Neurol. 2008;46 Suppl 1:S65-8. Spanish. PMID 18302126
- [Result] Rey Cao A, Canales Lacruz I, Taboas Pais MI. [Quality of life perceived by the elderly. Results of the "Memory in movement" program which provide cognitive stimulation using motricity]. Rev Esp Geriatr Gerontol. 2011 Mar-Apr;46(2):74-80. doi: 10.1016/j.regg.2010.08.005. Epub 2011 Mar 25. Spanish. PMID 21440332
- [Result] Wenisch E, Cantegreil-Kallen I, De Rotrou J, Garrigue P, Moulin F, Batouche F, Richard A, De Sant'Anna M, Rigaud AS. Cognitive stimulation intervention for elders with mild cognitive impairment compared with normal aged subjects: preliminary results. Aging Clin Exp Res. 2007 Aug;19(4):316-22. doi: 10.1007/BF03324708. PMID 17726363
- [Result] Jean L, Bergeron ME, Thivierge S, Simard M. Cognitive intervention programs for individuals with mild cognitive impairment: systematic review of the literature. Am J Geriatr Psychiatry. 2010 Apr;18(4):281-96. doi: 10.1097/JGP.0b013e3181c37ce9. PMID 20220584
- [Result] Novoa AM, Juarez O, Nebot M. [Review of the effectiveness of cognitive interventions in preventing cognitive deterioration in healthy elderly individuals]. Gac Sanit. 2008 Sep-Oct;22(5):474-82. doi: 10.1157/13126930. Spanish. PMID 19000530